CLINICAL TRIAL: NCT02043769
Title: Enhanced Surveillance and 2 Year Outcomes of Children Enrolled on Antiretroviral Therapy (ART) in Public Health Facilities in the Eastern Cape Province, South Africa
Brief Title: Pediatric Enhanced Surveillance Study
Acronym: PESS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Research Director, ICAP, Columbia University
Other Study IDs: AAAI1736; U2GPS001537 (NIH); U262PS223540 (Other Grant/Funding Number: MCAP)
Record Dates: First submitted 2014-01-13; First posted 2014-01-23 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Human Immunodeficiency Virus (HIV); Acquired Immune Deficiency Syndrome (AIDS)
Keywords: South Africa; Eastern Cape; Child ARV; CLWHIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Small amounts of additional blood will be drawn at the same time as routine blood draws and presents minimal risk to subjects (5cc of additional whole blood may be drawn from infants 1 month to 12 months of age or less than 10 kg in weight; 5 to 10 cc of additional blood may be drawn from children older than 12 months of age or >10 kg in weight); these risks usually include bruising at the site of the venipuncture, transient pain and a negligible chance for infection. No more than three attempts to obtain the blood specimens will be allowed per patient per blood collection visit. If collection of a blood sample/s fails this may be attempted at the next scheduled visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective Cohort: The prospective cohort surveillance will be built upon and support the routine clinical care, visit schedule and monitoring system at each study site. Eligible HIV-infected ART naïve children who are accessing care at study sites will be recruited sequentially for study enrollment. Children enrolled in the surveillance study will attend study visits co-scheduled to coincide with routine clinical visits. Study nurses will:
  1. review routinely collected information;
  2. conduct questionnaires with caregiver and child;
  3. conduct additional assessments of child;
  4. contact the caregiver by phone or through home visits for active follow-up for up to 24 months; and
  5. conduct active follow-up including appointment reminders by means of phone calls and defaulter tracking.

SUMMARY:
The Pediatric Enhanced Surveillance Study is a three part study of HIV-infected infants and children in South Africa to examine, clinical, immunologic, virologic, metabolic, psychosocial and behavioral outcomes. This study has two parts: (1) comprehensive de-identiﬁed records review of all HIV-infected children enrolled in at the pediatric Wellness and ART clinics at the ﬁve study sites; and (2) a prospective cohort surveillance study with active consented enrollment with 12-24 months of follow-up. As part of the prospective cohort, the study will aim to collect outcomes on children lost to follow-up, including causes of death through review of death certiﬁcates in the clinical chart and through verbal autopsy reports. The study will provide insights into overall outcomes for the larger pediatric patient populations in the province and South Africa. This work is designed in collaboration with the provincial health authorities of the Eastern Cape Department of Health (EC), The International Center for acquired immune deficiency syndrome (AIDS) Care and Treatment Programs (ICAP) South Africa and Center of Disease Control (CDC)-South Africa in support of the South African National ART Program for Children and aims to collect and analyze accurate, relevant and useful information that will be available on children seen at facilities. For the prospective cohort study, we will aim to enroll 400 children newly initiated on ART at 5 health facilities in the Eastern Cape of South Africa who will be actively followed for up to 24 months.

DETAILED DESCRIPTION:
South Africa is one of the countries hardest hit by the HIV/AIDS epidemic. There are more than 5 million people living with HIV in South Africa, including 280,000 children under the age of 15. Most HIV positive children acquire infection through mother-to-child transmission; in South Africa 29.3% of pregnant women attending antenatal services are HIV-infected. Furthermore, it is estimated that HIV is the cause of 35% of all deaths in children under five in South Africa. The South African government began a national rollout of HIV treatment for adults and children in 2003. As of 2007, an estimated 32,060 children under the age of 15 were receiving antiretroviral therapy (roughly 30% of those in need). There is an urgent need to obtain more comprehensive, in-depth, profiles of children enrolled in HIV care with a focus on documenting outcomes, particularly timing and causes of death, reasons for loss to follow-up, timing and frequency of treatment failure, adverse events, metabolic complications and psychosocial aspects of HIV disease.

ELIGIBILITY:
Inclusion Criteria:

* The child is eligible for antiretroviral therapy (ART) initiation based on the South African Pediatric HIV guidelines.
* The child has documentation of being HIV-infected by a positive HIV-Deoxyribonucleic acid (DNA) polymerase chain reaction (PCR), detectable HIV ribonucleic acid (RNA) viral load or a positive HIV antibody test (>18 months of age).
* The child has no prior history of treatment with ART other than prophylaxis for preventing mother to child transmission (PMTCT) (may be initiating ART on day of enrollment in study).
* The child is between 1 month and 12 years of age.
* The parent or legal guardian provides written consent for participation.
* The child provides assent for participation based on South African guidance for minors.

Exclusion Criteria:

* Any subject not meeting all of the above inclusion criteria will not be eligible for the study.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Human immunodeficiency virus (HIV)-infected children accessing HIV care and treatment services in the Eastern Cape of South Africa are the population of interest for the overall study.
  * Records review: All children with a record of care at the study facilities in the Wellness or antiretroviral (ART) clinic will form the study population.
  * Prospective cohort: ART-naïve children receiving care at participating sites who have reached eligibility for ART and consent to participate will form the study population. The sample for the study will be a subset of all children enrolled and receiving care at these public health care facilities.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of children alive and in care at 12 and 24 months after treatment initiation | Up to 24 months
  We will measure the proportion of children alive and in care at 12 and 24 months after treatment initiation amount prospective cohort participants through routine clinical and study visits.

SECONDARY OUTCOMES:
Proportion of the children enrolled in human immunodeficiency virus (HIV) care and treatment services | Up to 24 months
  We will describe the proportion of the children enrolled in HIV care and treatment services at the study facilities who start treatment and are retained in care for 6, 12, 24, 36 and 48 months by reviewing clinical records at each facility.
Proportion of children lost to follow-up | Up to 24 months
  We will describe the proportion of children lost to follow-up after enrollment in care and in those starting treatment by reviewing clinical records of study participants.
Proportion of children with documented deaths | Up to 24 months
  We will describe proportion of children with documented deaths and causes of deaths and time to death (from enrollment) by reviewing clinical records of participants.
Proportion of children who are virologically suppressed | Up to 24 months
  We will measure the proportion of children who are virologically suppressed (< 400 copies/mL, per South African National Guidelines) at 12 and 24* months after treatment initiation in the prospective cohort through routine clinical and study visits.
Proportion of children on antiretroviral therapy (ART) with diminished CD4 (cluster of differentiation 4) counts | Up to 24 months
  We will measure the proportion of children, aged 2 to 5 years, on ART with CD4% <10% at 12, 24* months after treatment initiation and children older than 5 years on ART with CD4 count of < 100 at 12, 24 months after treatment initiation. These outcomes will be measured in participants of the prospective cohort who will give additional blood samples during routine clinical care.
Proportion of children on antiretroviral therapy (ART) progressing to WHO Stage 4 disease | Up to 24 months
  We will measure the proportion of children on ART progressing to WHO Stage 4 disease at 12 and 24 months after treatment initiation in the prospective cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Abrams, MD, Principal Investigator — ICAP-NY, Columbia University
Locations (5):
- South Africa (5):
  - Cecilia Makiwane Hospital, East London, Amathole
  - Frere Hospital, East London, Amathole
  - Dora Ngiza Hospital, Port Elizabeth, Nelson Mandela Bay
  - Kwazakhele Community Health Center, Port Elizabeth, Nelson Mandela Bay
  - Motherwell Community Health Center, Port Elizabeth, Nelson Mandela Bay